CLINICAL TRIAL: NCT07292350
Title: Investigation of the Effects of a Neuromuscular Control-Focused Posture Training Program on Neck and Upper Back Muscle Activation in Butchers: A Randomized Controlled Trial
Brief Title: Investigation of the Effects of a Neuromuscular Control-Focused Posture Training Program in Butchers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Assoc.Prof.Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar78
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Work-related Illness; Neck Pain; Back Pain
MeSH Terms: conditions — Neck Pain; Back Pain | interventions — Ergonomics; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): only those who received ergonomics training
  Interventions: Other: ergonomics training
- exercise (Experimental): those who received exercise along with ergonomics training
  Interventions: Other: ergonomics training; Other: ergonomics training + exercise

INTERVENTIONS:
Other: ergonomics training — Each of the control group participants will receive separate ergonomics training. The content of this training will include the topics of "what is ergonomics, the purpose of ergonomics, musculoskeletal diseases in employees, work-related musculoskeletal risk factors
Other: ergonomics training + exercise — * Deep cervical flexor activation
  * Chin-tuck
  * 2-3 cm head lift endurance training
  * Scapular stabilization exercises
  * Retraction + depression
  * Serratus Anterior activation
  * Punch progressions in the supine position
  * Pectoral and upper trapezius stretching exercises
  * Functional posture training
  * Correction of butchers' forward bending and rotation movements when using knives
  * Ergonomic posture control during the task
  Arms: exercise

SUMMARY:
The aim of this study was to evaluate the effect of a neuromuscular posture training program implemented in butchers on neck pain, posture quality and upper back muscle control.

DETAILED DESCRIPTION:
The study population consists of butchers in Istanbul. Butchers will be included in the study after obtaining their informed consent. Participants will be randomized and divided into two equal groups. These groups will be designated as exercise and control groups. All participants will receive ergonomic training, while those in the exercise group will additionally receive neuromuscular exercises. At the beginning and end of the study, all participants will be assessed using the Visual Analog Scale, Neck Disability Index, Deep Cervical Flexor Endurance Test, Lateral Scapular Slide Test, Disabilities of the Arm, Shoulder, and Hand - Short Version, and Pittsburgh Sleep Quality Index.

ELIGIBILITY:
Inclusion Criteria

* Being over 18 years of age
* Actively working as a butcher in Istanbul
* Actively participating in the profession for at least 5 years
* Not having experienced acute trauma to the neck or back region within the last 3 months
* Being physically capable of participating in neuromuscular posture training
* Signing the Informed Voluntary Consent Form

Exclusion Criteria

Persons with the following characteristics will not be included in the study:

* Being under 18 years of age
* Not actively practicing butchery
* Having undergone surgery to the neck, spine, or shoulder region within the last 6 months
* Serious neurological conditions such as acute cervical disc herniation, radiculopathy, or myelopathy
* Systemic diseases such as cancer or serious cardiovascular disease
* Severe balance disorder/vestibular disorder
* Health condition that would prevent the safe continuation of exercise practice

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 10 weeks
  This index evaluates sleep quality and disturbance over the past month. It contains a total of 24 questions. 19 of these questions are answered by the person's self-assessment, and 5 of them are answered by the roommate who shares the same room with the person. The 5 questions answered by the person's roommate are not included when calculating the score. In scoring, the lowest (0) and the highest (21) points are obtained. A score of 4 and above indicates poor sleep quality
Quick-Arm, Shoulder and Hand Disabilities Survey functional scale | 10 weeks
  The Quick Arm, Shoulder and Hand Disabilities Survey score is calculated as follows: At least 10 out of the 11 items must be answered. Each answered question will have a maximum value of 5. These values are then transformed into a score of 100 by subtracting 1 and multiplying by 25. This transformation is done to compare the scores with other scales ranging from 0 to 100. A high score indicates significant dysfunction.
  Quick Arm, Shoulder and Hand Disabilities Survey Score = [(Sum of responses / n) - 1] X 25 n: the number of questions answered.
Neck Pain Disability Index Questionnaire | 10 weeks
  The scale includes 10 titles. It includes pain sensitivity, heavy lifting, personal hygiene, reading, sleep, headache, concentration, work, driving, social activities. There are 6 answer options according to the severity of the limitation or pain. Scoring is between 0 and 5. The highest score is 50 and the least is 0. The neck disability level classification according to the total score is as follows 0-4: no restrictions 5-14: mild limitation 15-24: moderate limitation 25-34: severe limitation 34 and up: completely restricted

CONTACTS AND LOCATIONS:
Overall Officials: Esra Çal, Study Chair — Uskudar University
Locations (1):
- Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gur I, Sevgin O, Dikmen Hosbas B. Effectiveness of ergonomics training and exercise in tea workers: a randomized controlled trial. Int Arch Occup Environ Health. 2025 Dec;98(9-10):945-955. doi: 10.1007/s00420-025-02185-0. Epub 2025 Nov 18. PMID 41251731
- [Background] Zengi H, Safran EE, Sevgin O. The effect of home exercises with kinesiotaping on pain, functionality, and work performance in bus drivers with non-specific neck pain. J Back Musculoskelet Rehabil. 2024;37(6):1617-1630. doi: 10.3233/BMR-240001. PMID 38943382
- [Background] Pehlevan E, Sevgin O. Effect of exercise given to factory workers with ergonomics training on pain and functionality: A randomized controlled trial. Work. 2024;78(1):195-205. doi: 10.3233/WOR-230663. PMID 38701125